CLINICAL TRIAL: NCT02615704
Title: Evaluation of an Electronic Device Based Support Tool for ACS Patients: Brilique (Ticagrelor) Treatment Adherence (eMocial)
Brief Title: "Me and My Heart" Study
Acronym: eMocial
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5130C00161
Record Dates: First submitted 2015-11-11; First posted 2015-11-26 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Acute Coronary Syndrome
Keywords: Brilique treatment adherence via electronic device application (APP)
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Micro-Electrical-Mechanical Systems; Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Active APP with MEMS: ACS patients 18 years or older with access to an electronic device (compatible with the patient support tool), diagnosed with STEMI, NSTEMI or UA treated with twice daily Brilique(ticagrelor) co administered with low dose acetylsalicylic acid according to the prescription recommendation using active APP with MEMS
  Interventions: Device: Active group with MEMS
- Active APP without MEMs: ACS patients 18 years or older with access to an electronic device (compatible with the patient support tool), diagnosed with STEMI, NSTEMI or UA treated with twice daily Brilique(ticagrelor) co administered with low dose acetylsalicylic acid according to the prescription recommendation using active APP without MEMS
  Interventions: Device: Active group without MEMS
- Control APP with MEMS: ACS patients 18 years or older with access to an electronic device (compatible with the patient support tool), diagnosed with STEMI, NSTEMI or UA treated with twice daily Brilique(ticagrelor) co administered with low dose acetylsalicylic acid according to the prescription recommendation using control APP with MEMS
  Interventions: Device: Control group with MEMS
- Control APP without MEMS: ACS patients 18 years or older with access to an electronic device (compatible with the patient support tool), diagnosed with STEMI, NSTEMI or UA treated with twice daily Brilique(ticagrelor) co administered with low dose acetylsalicylic acid according to the prescription recommendation using control APP without MEMS
  Interventions: Device: Control group without MEMS

INTERVENTIONS:
Device: Active group with MEMS — Patients treated with twice daily Brilique (ticagrelor) co administered with low dose of acetylsalicylic acid with APP as support tool and with MEMS
  Other Names: Group A with MEMS
  Groups: Active APP with MEMS
Device: Active group without MEMS — Patients treated with twice daily Brilique (ticagrelor) co administered with low dose of acetylsalicylic acid with APP as support tool but without MEMS
  Other Names: Group A without MEMS
  Groups: Active APP without MEMs
Device: Control group with MEMS — Patients treated with twice daily Brilique (ticagrelor) co administered with low dose of acetylsalicylic acid without APP as support tool but with MEMS
  Other Names: Group B with MEMS
  Groups: Control APP with MEMS
Device: Control group without MEMS — Patients treated with twice daily Brilique (ticagrelor) co administered with low dose of acetylsalicylic acid without APP as support tool and without MEMS
  Other Names: Group B without MEMS
  Groups: Control APP without MEMS

SUMMARY:
An electronic device application (APP) "Mein Herz und ich" has been developed specifically for acute coronary syndrome (ACS) patients who are prescribed to Brilique (ticagrelor) to increase adherence to treatment (medication and lifestyle changes) by a combination of reminders on medication intake, information on the importance of treatment, motivation by supportive messages, and visualisation of individual lifestyle choices' effect on cardiovascular risk. The aim of this study is to evaluate the effectiveness of this patient support tool

DETAILED DESCRIPTION:
The target population are patients hospitalised with acute coronary syndrome (ACS) 18 years or older with access to an electronic device (compatible with the patient support tool), diagnosed with ST elevation myocardial infarction (STEMI), non-ST elevation myocardial infarction (NSTEMI), unstable angina pectoris (UA) and treated with twice daily Brilique (ticagrelor) co administered with low dose acetylsalicylic acid (ASA) according to the prescription recommendation, within 14 days following the diagnosis of the ACS event. Patients will be randomised 1:1 into an active group receiving the patient support tool under investigation via electronic device application (APP) and a control group without patient support tool. In addition, both active and control group will be randomised 1:1 to a group with or without use of a Medical Event Monitoring System (MEMS) for evaluation of treatment adherence. Patient questionnaires for evaluation of lifestyle changes, and quality of life will be administered at the beginning (Visit 1) and end (Visit 2) of the observation period. In addition, questionnaires for adherence, treatment attitudes, health care utilization and risk factors will be administered in monthly intervals

This is a randomised investigation according to paragraph 23b of the German Medical Device Law examining the impact of the APP use on drug adherence, drug persistence and lifestyle changes in patients who have been prescribed Brilique (ticagrelor) as part of normal clinical practice in a 12 month timeframe after their ACS episode.

The device has a European Conformity Declaration (CE-mark). In this study no investigational product will be dispensed to the study participants. Patients will need to provide their own Brilique(ticagrelor) supply from the pharmacy, as in common clinical practice. Further, assessments in this study will not be used for guiding the treatment of the patients participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated patient informed consent prior to randomisation
* Female or male aged 18 years or older
* Acute Coronary Syndrome patients, diagnosed with ST elevation myocardial infarction, non-ST elevation myocardial infarction or unstable angina pectoris treated with Brilique (ticagrelor) prior to inclusion into this study and for whom the treating physician intends to continue prescribing twice daily Brilique (ticagrelor) co administered with low dose acetylsalicylic acid according to the prescription recommendation, within 14 days following the diagnosis of the ACS event
* Ability to read, understand and write German
* Patients must have access to an electronic device (compatible with the patient support tool) and willing to use it on a daily basis

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff and/or staff at the study site and application developer)
* Participation in another clinical study with an investigational product or medical device during the last 30 days, excluding prospective/retrospective register based studies that do not require any extra visits in addition to ordinary health care
* Patients on treatment with Oral Anti-Platelet drugs other than Brilique (ticagrelor)
* Patients with contraindication to the use of Brilique (ticagrelor)
* Patients accepted/with a plan for thoracic surgery (coronary artery bypass grafting, CABG) or any other elective surgery that cannot be postponed until after study participation
* Presence of serious/severe co-morbidities in the opinion of the Investigator which may limit life expectancy (<1 year)
* For women only: patients who are currently pregnant (confirmed with positive pregnancy test) or breast feeding

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population are acute coronary syndrome (ACS) patients 18 years or older with access to an electronic device (compatible with the patient support tool), diagnosed with ST elevation myocardial infarction, non-ST elevation myocardial infarction or unstable angina pectoris treated with twice daily Brilique (ticagrelor) co administered with low dose acetylsalicylic acid according to the prescription recommendation, within 14 days following the diagnosis of the ACS event.
Sampling Method: Non-Probability Sample
Enrollment: 677 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Percentage of tablets taken during the observation phase | An average of 48 weeks
  Adherence to prescribed treatment according to questions 1-4 in the Brilique Adherence Questionnaire (BAQ) including a scoring system for quantification from 0-14 (i.e. one deduction for every missed Brilique (ticagrelor) tablet per week with 7 days and twice daily dosing). The BAQ will be delivered via the APP every 4 weeks. The percent of tablets taken from the last week asked for in BAQ, will be representing the last 4 weeks of Brilique use.

SECONDARY OUTCOMES:
Percentage of tablets taken during the observation phase | An average of 48 weeks
  Tablets taken measured by a Medical Event Monitoring System (MEMS) to record a time stamp for every tablets taken
The percent change in key risk factors | 1 year
  Key risk factors like blood pressure, laboratory parameters (if available: LDL cholesterol, HDL cholesterol, HbA1c, body weight, and BMI)
Change in Quality of Life | 1 year
  Change in Quality of Life assessed by Short Form 36 Questionnaire (SF-36v2)
Change in patient reported lifestyle changes | An average of one year
  Lifestyle changes assessed by a Lifestyle Changes Questionnaire (LSQ) at V1 and V2 (patient reported outcome (PRO) instrument
Disease understanding and treatment awareness | Every four weeks during 48 weeks observational phase
  Assessed according to questions 5-11 in the BAQ
Health care utilization | Every four weeks during the 48 weeks observational phase
  Assessed on the questions 12-15 in the BAQ

OTHER OUTCOMES:
Cardiovascular risk score GRACE 2.0 | During baseline
  Impact of GRACE 2.0 risk score at baseline on adherence as assessed by BAQ
Treatment gaps according to missed tablets obtained in the subgroup of patients equipped | During 48 weeks observational phase
  Missed tablets (based on MEMS) compared between randomized groups
Patients' report on the use of alternative medication reminder or other health APPs | An average of one year
  Usage of other medication reminder or health apps
For the active treatment group, data on the use of the patient support tool | An average of one year
  The number of times the APP is used during the study through an analysis of the recorded user data
For the active treatment group, responses to the questions of the System Usability Scale (SUS) | An average of one year
  Assessment of SUS replies at visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Florian Krackhardt, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (29):
- Germany (29):
  - Research Site, Bad Berka
  - Research Site, Bad Bevensen
  - Research Site, Bad Krozingen
  - Research Site, Barby
  - Research Site, Berlin
  - Research Site, Bernau
  - Research Site, Chemnitz
  - Research Site, Coburg
  - Research Site, Düsseldorf
  - Research Site, Erkrath
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Gelsenkirchen
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Kleve
  - Research Site, Lübeck
  - Research Site, Mainz
  - Research Site, Mönchengladbach
  - Research Site, Münster
  - Research Site, Oldenburg
  - Research Site, Regensburg
  - Research Site, Rostock
  - Research Site, Rotenburg (Wümme)
  - Research Site, Siegen
  - Research Site, Tegel
  - Research Site, Wuppertal

REFERENCES:
- [Derived] Krackhardt F, Jornten-Karlsson M, Waliszewski M, Knutsson M, Niklasson A, Appel KF, Degenhardt R, Ghanem A, Kohler T, Ohlow MA, Tschope C, Theres H, Vom Dahl J, Karlson BW, Maier LS. Results from the "Me & My Heart" (eMocial) Study: a Randomized Evaluation of a New Smartphone-Based Support Tool to Increase Therapy Adherence of Patients with Acute Coronary Syndrome. Cardiovasc Drugs Ther. 2023 Aug;37(4):729-741. doi: 10.1007/s10557-022-07331-1. Epub 2022 Apr 20. PMID 35441926
- [Derived] Krackhardt F, Maier LS, Appel KF, Kohler T, Ghanem A, Tschoepe C, Dahl JV, Degenhardt R, Niklasson A, Ahlqvist M, Waliszewski MW, Jornten-Karlsson M. Design and rationale for the "Me & My Heart" (eMocial) study: A randomized evaluation of a new smartphone-based support tool to increase therapy adherence of patients with acute coronary syndrome. Clin Cardiol. 2019 Nov;42(11):1054-1062. doi: 10.1002/clc.23254. Epub 2019 Sep 6. PMID 31490566
- See also: D5130C00161 CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5130C00161&attachmentIdentifier=045cad0f-df85-4051-aafb-dd74c86358a0&fileName=D5130C00161_CSR_Synopsis_Redacted.pdf&versionIdentifier=